CLINICAL TRIAL: NCT00631020
Title: Determining the Efficacy of Cognitive-behavioral Motivational Enhancement +/- Nicotine Replacement Therapy for Adolescents
Brief Title: Youth Smoking Cessation: Therapy +/- "The Patch"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Philip Morris USA (Unknown)
Responsible Party: Principal Investigator, Steve Shoptaw, Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PM 20063287
Record Dates: First submitted 2008-02-27; First posted 2008-03-07 (Estimated); Results first posted 2015-04-22 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Smoking
Keywords: Youth; Smoking; Tobacco; Adolescent; Dependence; Teen smoking; Smoking and youth; Youth and tobacco
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBME +/- NRT (Experimental): 6 weeks CBME with optional 4 weeks NRT
  Interventions: Behavioral: CBME; Drug: Optional NRT

INTERVENTIONS:
Behavioral: CBME — 6 weeks of once a week one-on-one CBME
Drug: Optional NRT — NicoDerm CQ nicotine transdermal patch

SUMMARY:
Reducing tobacco use by adolescents is a national health priority. In recent polls, most adolescent smokers reported having tried unsuccessfully to quit. Smoking cessation treatment during adolescence has the potential to interrupt the progression to nicotine dependence, which is attended by a wide range of negative health consequences. Given the need for effective smoking cessation programs aimed at youth, scientifically rigorous research is warranted to reduce adolescent smoking. This project will address gaps in the scientific treatment literature. The goal of this project is to develop a tailored, practical, and efficacious smoking cessation intervention. Combined with other efforts in the field, this work can provide an initial guide to an evidence-based treatment for smoking cessation in youth.

In keeping with developments in other fields of medicine, we believe that further advances in smoking cessation will move towards a goal of personalized treatment. Such an individualized approach for adolescent smoking cessation will be informed by further investigation of the relationships between outcomes in this trial. To serve these goals, we propose the following program:

Youths who smoke regularly will receive a 6 week intervention using "cognitive-behavioral motivational enhancement" (CBME) supplemented by nicotine replacement therapy (NRT), if youth and parents desire this option. Furthermore, youth has to smoke more than 5 cigarettes a day in order to qualify for nicotine replacement therapy. This approach is consistent with treatment guidelines for smoking cessation (Fiore 2000).

Compared with participants who fail to achieve smoking cessation, those who successfully achieve smoking abstinence during intervention, will have lower baseline rates of comorbid ADHD, lower depressive symptom scores, enhanced readiness to quit, more negative attitudes towards smoking, fewer friends who smoke, and fewer family members who smoke. The investigators predict that the intervention will help youth to quit smoking and will examine predictions of successful quitting.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable cause of death in the United States, and current estimates project that 6.4 million of our nation's youth will die prematurely from a smoking-related disease (Fellows et al., 2002). Extant data suggest that three of every five adolescent smokers are nicotine-dependent, and that some subgroups of adolescents are at higher risk for dependence (e.g., daily or heavy smokers, incarcerated youth, youth in vocational schools, depressed youth, youth with Attention Deficit Hyperactivity Disorder (ADHD)). Adolescent tobacco smoking increases risk for a wide range of negative health consequences (Abrantes et al., 2005; Anda et al., 1990; Biederman et al., 2006; Escobedo et al., 1998; Kandel et al., 1986; Kollins et al., 2005; Wilens & Dodson 2004). For example, smoking-related cancer risk is increased with early age of initiating smoking and longer time of smoking, underscoring the importance of addressing this health risk behavior in youth (Centers for Disease Control and Prevention, 1994).

Reducing tobacco use by adolescents is a national health priority (see Healthy People 2010, Objective, 27.2 (Office of Disease Prevention and Health Promotion 2000)). Approximately 4% of 8th graders, 7.5% of 10th graders, and 13.6% of 12th graders smoke daily and almost half of these youths smoke ≥ half a pack per day (Johnston & O'Coner 2005). In recent polls, most adolescent smokers reported having tried unsuccessfully to quit (Grimshaw et al., 2003; Hollis et al., 2003). Smoking cessation treatment during adolescence has the potential to interrupt the progression to nicotine dependence, which is attended by a wide range of negative health consequences (Anda et al., 1990; Escobedo et al., 1998; Kandel & Davies 1986). Given the need for effective smoking cessation programs aimed at youth, scientifically rigorous research is warranted to reduce adolescent smoking (Backinger et al., 2003). This project will address gaps in the scientific treatment literature.

In keeping with developments in other fields of medicine, we believe that further advances in smoking cessation will move towards a goal of personalized treatment. In order to optimize the aim for personalized treatment we will include genetic testing. For some smoking cessation treatments, evidence has begun to accumulate that the inter-individual variability in response to treatment benefits and side effects may be influenced by inheritance. In the smoking cessation treatment literature, some observations have already been made suggesting that common gene variants may be associated with different treatment outcomes. The association between depression and smoking has led to interest in whether the short allele of the serotonin transporter gene may be associated with increased vulnerability to smoking and nicotine dependence, although to our knowledge this has yet to be demonstrated (Brody, et al. 2005). Such findings suggest that individual vulnerability to the reinforcing effects of smoking, and most important to this study differences in quitting success, could be partially predicted by individual genotype. Additionally, motivational and psychosocial factors have also been identified as likely predictors of treatment response. We are seeking predictors that would allow us to reach the ultimate objective: to contribute to an algorithm to better match youth and effective smoking cessation treatment.

Specific Aims of the study are as follows:

1. To evaluate an intervention for adolescent smoking cessation.
2. To examine moderators and mediators of successful smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following inclusion criteria:

* age of 14-21 years, inclusive
* regular cigarette smoking at least five times a day in the month before entry into the study and initiation of smoking at least 6 months before entry
* A score of 35 or greater on the Cigarette Dependence Scale-12
* youth provide informed assent (for youth <18 yr) or consent (for youth ≥18 yr) and parents provide informed consent to participate in the project
* documented approval to participate from the participant's treating physician for participants currently receiving treatment for a serious medical or psychiatric condition
* current contact information (address, telephone number), which is needed for follow-up
* able to complete study assessments and participate in the intervention (e.g., lives < 1 hr. away from the site, has family to participate in the intervention, does not have mental retardation)
* youth or primary caregivers speak English or Spanish

Exclusion Criteria:

Participants must meet none of the following exclusion criteria in order to be eligible to receive optional nicotine replacement:

* smoke less than 5 cigarettes per day
* have serious cardiovascular disease, including uncontrolled hypertension, coronary artery disease, serious cardiac arrhythmias, vasospastic disease, or angina, due to potential cardiovascular effects of nicotine, as determined via the baseline medical history and physical exam
* have a medical condition that could be made worse by treatment with nicotine, including poorly controlled insulin dependent diabetes, uncontrolled hyperthyroidism, pheochromocytoma, severe oropharyngeal, esophageal, or peptic ulcer disease, or severe renal or hepatic impairment as determined via the baseline medical history and physical exam
* have an allergy to adhesive tape or latex or serious dermatologic disease (excluding minor skin conditions such as mild eczema) due to potential for skin allergy to patch
* have a known allergy to nicotine or any component of the nicotine patches
* be receiving treatment with adenosine or bupropion due to potential drug-drug interactions
* be pregnant or sexually active and not using reliable birth control methods consistently (for females)

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2007-12; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Shoptaw, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- CBME +/- NRT: 6 weeks CBME with optional NRT for 4 weeks
Period: Overall Study
Arm/Group | CBME +/- NRT
Started | 34
Completed | 26
Not Completed | 8
Not completed — Lost to Follow-up | 7
Not completed — Incarcerated | 1

BASELINE CHARACTERISTICS:
Groups:
- CBME +/- NRT: 6 weeks of once a week CBME with optional 4 weeks NRT
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 19 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Acceptance of Nicotine Replacement Therapy
Description: Participants were offered optional nicotine replacement therapy (NRT). The number of participants that opted for NRT was measured.
Time Frame: week 2
Measure: Number; unit: participants
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 34
participants | 26

2. Primary Outcome: Retention in Trial
Description: Retention in trial is defined as completing the 6-week intervention (attended week6, yes/no)
Time Frame: week 6
Measure: Number; unit: participants
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 34
participants | 26

3. Primary Outcome: 7-day Smoking Abstinence at End of Treatment (Week 6) and at Follow-up Visits (Weeks 12, 16, 24)
Description: The primary index of smoking behavior will be subject's self-report of smoking using a diary method for the past 7 days prior to the assessment. The subject self-report will be supplemented by: expired CO and by urine cotinine concentrations. Abstinence (yes/no) will be defined as no cigarettes during the past 7 days and an expired CO of <=8 ppm.
Time Frame: week 6, 12, 16 and 24
Measure: Number; unit: participants
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 26
participants
  Week 6 (n=26) | 8
  Week 12 (n=25) | 6
  Week 16 (n=23) | 4
  Week 24 (n=23) | 2

4. Secondary Outcome: Changes in Tobacco Withdrawal Symptoms Compared to Baseline
Description: Tobacco withdrawal symptoms were measured using the Minnesota Nicotine Withdrawal Scale (MNWS). Eight withdrawal symptoms are each rated for their severity on a scale from 0 (not present) to 4 (severe) for the past week and summed to calculate a total score at each time point, with a score range of 0-32. The average change from baseline for all participants at the specified time points were determined.
Time Frame: Weeks 6, 12, 16 and 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 26
units on a scale
  Week 6 (n=26) | -5.6 (7.3)
  Week 12 (n=25) | -5.7 (6.6)
  Week 16 (n=23) | -3.5 (6.8)
  Week 24 (n=23) | -4.3 (5.3)

5. Secondary Outcome: Change in Tobacco Dependence Compared to Baseline
Description: Tobacco dependence was measured using the Cigarette Dependence Scale (CDS-12). The CDS-12 scale is a 12-item scale that assesses some components of formal diagnostic systems' (e.g., DSM-IV and ICD-10) definitions of dependence with an emphasis on compulsion to smoke, withdrawal, loss of control, time allocation, neglect of other activities, and persistence despite harm. Response choices are on a five-point Likert scale to measure dependence (low =1; high = 5), the total score is the sum of all 12 items with a score range of 12 - 60. The change in scores from baseline at each time point were measured.
Time Frame: Weeks 6, 12, 16 and 24
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 26
units on a scale
  Week 6 (n=26) | -19 (12)
  Week 12 (n=25) | -14.3 (12.9)
  Week 16 (n=23) | -12.2 (13)
  Week 24 (n=23) | -8.8 (14.3)

6. Secondary Outcome: Change in Number of Cigarettes/Day During the Past 7-days Compared to Baseline
Description: Change from baseline self report of number of cigarettes per day compared to the past 7 days at each time point.
Time Frame: Weeks 6, 12, 16 and 24
Measure: Mean (Standard Deviation); unit: cigarettes/day
Arm/Group | CBME +/- NRT
Number analyzed (Participants) | 26
cigarettes/day
  Week 6 (n=26) | 3.1 (4.6)
  Week 12 (n=25) | 3.9 (4.2)
  Week 16 (n=23) | 3.4 (4.2)
  Week 24 (n=23) | 6.7 (6.2)

ADVERSE EVENTS:
Description: As a safety measure, participants will consult with the study physician or licensed nurse practitioner once a week about their general health. Any physical or clinical change or illness, whether or not it is considered study drug related, will be recorded on the medical record chart and adverse event case report form.
Arm/Group | CBME +/- NRT
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 20/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBME +/- NRT (N=34)
Rash-like reaction (Skin and subcutaneous tissue disorders) | 7 (10)
Insomnia (Psychiatric disorders) | 6 (7)
Craving (Psychiatric disorders) | 4 (6)
Nausea (Gastrointestinal disorders) | 3 (6)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Headache (Nervous system disorders) | 4 (4)
Irritable (Psychiatric disorders) | 4 (4)
Cold symptoms (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Anhedonia (Psychiatric disorders) | 1 (1)
Decreased concentration (Psychiatric disorders) | 1 (1)
Decreased energy (General disorders) | 1 (1)
Dental pain (Gastrointestinal disorders) | 1 (1)
Dizzy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Indigestion (Gastrointestinal disorders) | 1 (1)
Shaky (Psychiatric disorders) | 1 (1)
Strep throat (Infections and infestations) | 1 (1)
Stress (Psychiatric disorders) | 1 (1)
Toe pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tonsillar abscess (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Vivid dreams (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No